CLINICAL TRIAL: NCT04319042
Title: Influence of the Implant Loading Protocol on Implant Survival in Early Placed Single-tooth Implants in Mandibular First Molar Sites Using Computer-assisted Implant Surgery: A Randomized Clinical Trial (RCT).
Brief Title: Effect of Placing the Implant Crown on the Implant on the Same Day as the Implant vs. 4 Weeks Later.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITI 1455_2019
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Lower Molar Requiring Extraction
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Loading (Active Comparator): Group A. The implant receives an artificial tooth the same day as it is placed.
  Interventions: Procedure: Immediate Loading
- Early Loading (Active Comparator): Group B. The implant receives an artificial tooth 4 weeks after placement.
  Interventions: Procedure: Early Loading

INTERVENTIONS:
Procedure: Immediate Loading — The implant receives an artificial tooth the same day as it is placed.
  Arms: Immediate Loading
Procedure: Early Loading — The implant receives an artificial tooth 4 weeks after placement.
  Arms: Early Loading

SUMMARY:
In this study, participants with one lower first molar that require removal and replacement using dental implants will be enrolled. The implant will be inserted 12-16 weeks after tooth extraction and restored either immediately with an artificial tooth (fixed implant crown) in 50% of the cases or 4 weeks later in the remainder 50%. Immediate and early loading will be compared and the investigators expect no difference in terms of implant success and health of the tissue around the implant.

DETAILED DESCRIPTION:
Background

Dental implants placed between 12 and 16 weeks after tooth loss are a well-documented treatment option. Placing the artificial tooth (implant crown) on the implant the same day (immediate loading) or approximately 4 weeks after implant placement (early loading) are also treatment options with good scientific documentation. Computer-assisted implant surgery (sCAIS) and modern implant materials/surfaces increase treatment predictability and success in this context.

Clinical relevance

The timing of implant placement post-extraction and subsequent implant loading cannot be separated in modern implant therapy any longer. At the "Sixth ITI Consensus Conference" in Amsterdam, it was concluded that the clinical evidence and documentation of early implant placement combined with immediate or early implant loading in partially edentulous patients is currently insufficiently documented. However, this treatment protocol seems to be widely applied in daily practice. The planned study is designed to provide evidence for the application of early implant placement with partial bone-healing and either an immediate or an early loading protocol.

Hypothesis/Specific aims

H0: "Early placed single tooth implants by means of static computer-assisted implant surgery (sCAIS) in mandibular first molar sites with immediately loaded provisionals, show a survival rate comparable to early placed implants with an early loading protocol." Secondary parameters to be evaluated will be the prosthetic survival/ success, patient-centered outcomes (PROs), clinical peri-implant conditions, bone-level changes, alteration of peri-implant soft-tissue dimensions and the accuracy of digital implant planning.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years
* Willingness to sign informed consent and to participate in the study
* Plaque index according to Silness and Loe of < 35% [26]
* Presence of a mandibular first molar that has to be extracted
* Sufficient vertical interocclusal space for the placement of an implant crown (7 mm)
* Presence of an opposing natural or artificial tooth
* Ridge height sufficient for the placement of a ≥ 10 mm-long implant
* Sufficient ridge width for the placement of a 4.1mm diameter implant

Exclusion Criteria:

* Any physical or mental disorder that would interfere with the ability to perform adequate oral hygiene or the capability of providing written informed consent and compliance to the protocol
* Any disorder that would interfere with wound healing or represent a contraindication for implant surgery such as, but not limited to, uncontrolled diabetes or conditions resulting in or requiring immunosuppression, radiation, chemotherapy, frequent use of antibiotics or antiresorptive medication such as bisphosphonates
* Pregnancy or lactation
* Intention to become pregnant between inclusion and implant loading
* Heavy smoking habit with ≥ 10 cig/d
* Severe bruxism or clenching habits, present oro-facial pain
* Insufficient ridge width/height for the study implant
* Defect of any alveolar wall (secondary exclusion criterion at tooth extraction)
* ISQ < 70 (secondary exclusion criterion for Group A at implant placement, for Group B at loading visit)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2033-05 (Estimated)

PRIMARY OUTCOMES:
Implant Survival | 12 months
  Number of implants from both groups (i.e. immediate loading vs. early loading) fulfilling the criteria of survival and success after 12 months. The criteria are:
  * Absence of persisting subjective discomfort such as pain, foreign body perception and or dysaesthesia (e. g. painful sensation)
  * Absence of a recurrent peri-implant infection with suppuration (where an infection is termed recurrent if observed at two or more follow-up visits after the treatment with systemic antibiotics)
  * Absence of implant mobility on manual palpation
  * Absence of any continuous peri-implant radiolucency

SECONDARY OUTCOMES:
Prosthetic Success | 10 years
  Esthetics and correct function of the implant prosthetic will be analyzed by means of palpation, inspection and probing. Any prosthetic complication, e.g. chipping, screw loosening will be recorded.
Patient's satisfaction | 10 years
  Patient's satisfaction with the treatment result will be analyzed by means of questions (both oral and written, using validated questionnaires)
Clinical peri-implant soft tissue dimensions | 10 years
  Probing depth of the soft tissue surrounding the implant will be assessed using palpation, inspection and a periodontal probe.
Crestal bone level | 10 years
  Crestal bone-level changes will be assessed in the follow-up radiographs that are taken routinely after any implant treatment, using a dedicated imaging software.
Accuracy of digital implant planning | 12 months
  The difference between digitally planned and real/final implant position will be analyzed by superimposing the digitized final impression and the digital preoperative planning with the dedicated software. No additional exposure to radiation or additional impressions will be necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Simone FM Janner, PD Dr., Principal Investigator — University of Bern; Samir Abou-Ayash, Dr.med.dent., Principal Investigator — University of Bern
Locations (2):
- Switzerland (2):
  - Klinik für Oralchirurgie und Stomatologie, Bern
  - Klinik für rekonstruktive Zahnmedizin und Gerodontologie, Bern

IPD SHARING:
Plan to Share IPD: No